CLINICAL TRIAL: NCT00358189
Title: Deep Brain Stimulation and Motor Function in Parkinson's Patients
Brief Title: Effects of Deep Brain Stimulation for the Treatment of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B4061I
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2006-07

CONDITIONS: Parkinson
Keywords: deep brain stimulation; gait; manual dexterity; parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Deep Brain Stimulation

SUMMARY:
The purpose of this study is to assess the effects of unilateral deep brain stimulation on upper and lower extremity motor function in advanced Parkinson's disease patients. It is hypothesized the unilateral stimulation will lead to improvements in bilateral motor functioning.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic progressive degenerative illness in which dopaminergic neurons in the substantia nigra pars compacta deteriorate resulting in a reduction in striatal dopamine. Decreased levels of dopamine in PD patients results in varying combinations of akinesia, bradykinesia, tremor, rigidity and gait\postural instability. Parkinson's disease is the second most common neurodegenerative disorder, affecting nearly 1.2 million Americans with annual treatment costs approaching $25 billion. Deep brain stimulation (DBS) is a surgical approach developed for the treatment of advanced PD that provides promise in alleviating its motor deficits. The most common stimulation site for the treatment of advanced PD is the subthalamic nucleus (STN). Nearly 90 percent of patients involved in a multi-center trial with STN stimulation underwent single session bilateral implantation. It is generally accepted that bilateral STN stimulation improves upper and lower extremity function. However, bilateral STN stimulation may be associated with postoperative morbidity including cognitive deficits and neuropsychiatric changes. In contrast, the effects of unilateral STN stimulation on bilateral upper and lower extremity motor function are poorly understood. The question of whether to proceed with bilateral or unilateral surgery is important, as a significant number of patients for whom surgery is a consideration have relative contraindications such as age greater than 70, cognitive decline, or other medical conditions that may prevent bilateral implantation. Considering the risks for bilateral implantation may be greater than unilateral procedures, it is necessary to determine if unilateral stimulation is an effective means of ameliorating PD symptoms. The primary aim of this collaborative project is to determine the effects of unilateral STN DBS on functional upper (manual dexterity) and lower (postural stability and gait initiation) extremity motor performance in Veterans with advanced PD. The results from these studies have the potential to impact the use of DBS in the treatment of advanced PD. Positive bilateral results with unilateral stimulation of STN may allow patients not currently considered eligible for bilateral implantation to be considered for unilateral procedures as a method of treating PD symptoms. Our general hypothesis is that unilateral STN DBS acts to override disrupted neural activity of the basal ganglia in one hemisphere. The resultant normalized basal ganglia output to the SMA then allows for improved planning and control of bilateral actions. Bilateral upper and lower extremity motor performance will be quantified in a group of advanced PD patients with unilateral STN DBS patients while "on" and "off" stimulation. It is hypothesized that unilateral STN DBS will result in bilateral improvements in upper and lower extremity motor function.

ELIGIBILITY:
Inclusion Criteria:

* a) Patients must have had the Deep Brain Stimulator implanted for at least six months prior to enrollment.
* Hoehn and Yahr stage III or worse when off stimulation and medication
* Intractable, disabling motor fluctuations, dyskinesias or freezing episodes
* Age between 30-75 years
* Normal cognition
* Demonstrated good response to levodopa. In order to exclude patients with Parkinson's plus (i.e. progressive supranuclear palsy, multiple system atrophy, striato-nigral degeneration, etc) all patients included in this study must have demonstrated a good response to levodopa, defined as demonstrating at least 30% improvement in parkinsonian motor signs, based on UPDRS motor examination subscore following the administration of levodopa during their screening neurological exam.
* Unsatisfactory clinical response to maximal medical management A stable and optimal medical regimen of antiparkinsonian drug therapy for at least three months prior to or after surgery

Exclusion Criteria:

* Clinically significant medical disease that would increase risk of developing pre- or postoperative complications (e.g. significant cardiac or pulmonary disease, uncontrolled hypertension).
* Evidence of secondary or atypical parkinsonism as suggested by:
* History of CVA's, exposure to toxins, neuroleptics or encephalitis
* Neurologic signs of upper motor neuron or cerebellar involvement, supranuclear gaze palsy or significant orthostatic hypertension
* Dementia as evidenced by impairment in two neuropsychological domains and impaired or borderline neuropsychological function in one additional domain
* Use of DBS for psychiatric disorder (obsessive compulsive or depression)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-10; Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay L Alberts, PhD, Principal Investigator — Investigator
Locations (1):
- Louis Stoke Cleveland VA Medical Center, Cleveland, Ohio, United States